CLINICAL TRIAL: NCT00591370
Title: Phase II Trial of Extended-Dosing Temozolomide in Patients With Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-138
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Results first posted 2015-01-22 (Estimated); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Melanoma
Keywords: Memorial Sloan-Kettering Cancer Center patients with measurable, unresectable stage; III or IV melanoma
MeSH Terms: conditions — Melanoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 - Temozolomide (TMZ) (Experimental)
  Interventions: Drug: Temozolomide (TMZ)

INTERVENTIONS:
Drug: Temozolomide (TMZ) — One group treatment study

SUMMARY:
Temozolomide (also known as TMZ) is a chemotherapy drug given by mouth. It is similar to DTIC, the only FDA-approved chemotherapy for melanoma, but because temozolomide is given by mouth, it can be given daily over a long period of time. We think that temozolomidemay work best if it is given every day for 6 weeks at a time. Temozolomide given by this extended schedule is experimental, although we have found that it is safe and can shrink melanoma in some patients.

One big advantage of TMZ is that it is given by mouth instead of by vein. This means that it can be given daily over a long period of time rather than off and on like DTIC. We think that TMZ may work better if it is given every day for 6 weeks. TMZ given by this extended schedule is experimental although we have found that TMZ given in this way is safe and can shrink melanoma in some patients. When extended dosing TMZ was given with either thalidomide or long-acting interferon-α, about 30% of patients had their tumors shrink. We think that this shrinkage was due mostly to the TMZ since neither thalidomide nor interferon-α alpha work in melanoma by themselves.

In this study, we will treat patients with TMZ alone using this extended dosing schedule to see how many patients experience tumor shrinkage.

We also want to learn more about which tumors are more likely to shrink from TMZ treatment. We will test samples of your tumor for whether or not a gene called MGMT has been turned on,

ELIGIBILITY:
Inclusion Criteria:

* Stage III (unresectable) or Stage IV melanoma from a cutaneous or an unknown primary.
* Histologic proof of melanoma reviewed and confirmed at MSKCC
* Measurable disease (RECIST criteria)
* No prior chemotherapy for melanoma. Prior interferon, interleukin-2 or vaccine therapy are allowed.
* No other concurrent chemotherapy, immunotherapy, or radiotherapy
* Karnofsky performance status ≥ 60
* Adequate organ function defined as follows: ANC > 1500, Platelets > 100,000, creatinine < 2, Alkaline Phosphatase, AST and total bilirubin < 1.5x upper limit of normal. For patients with suspected Gilbert's syndrome bilirubin will not be a requirement.
* Tumor tissue for MGMT promoter methylation analysis and/or IHC must be available. In most cases, this will be unstained slides from previously-obtained paraffin-embedded tumor material. If this is not available, patients must have an easily-accessable tumor for biopsy (e.g. skin or lymph node).

Exclusion Criteria:

* History of CNS metastases unless brain metastases have been resected and the patient has been free from CNS recurrence for 6 months.
* Uveal or mucosal melanoma primary
* Frequent vomiting or medical conditions that could interfere with oral medication intake
* Serious infection requiring antibiotics, or nonmalignant medical illnesses that are uncontrolled or whose control might be jeopardized by the complications of this therapy.
* History of HIV infection even if on HAART
* Immunosuppressive drugs
* High dose vitamins and herbs
* Other on-going investigational therapy, concurrent chemotherapy, immunotherapy or radiotherapy.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2005-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Chapman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual-01/12/2005 Protocol Closed to Accrual-11/27/2007 Primary Completion Date-06/10/2008 Recruitment Location is the medical clinic
Groups:
- Temozolomide (TMZ): Temozolomide (TMZ) 75 mg/m2/day x 6 weeks every 8 weeks
Period: Overall Study
Arm/Group | Temozolomide (TMZ)
Started | 51
Completed | 49
Not Completed | 2
Not completed — Not Treated | 2

BASELINE CHARACTERISTICS:
Arm/Group | Temozolomide (TMZ)
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 23
  >=65 years | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 33
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Determine the Overall Objective Response Rate (CR and PR).
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: From start of treatment through 24 weeks after ending treatment
Measure: Number; unit: participants
Arm/Group | Temozolomide (TMZ)
Number analyzed (Participants) | 49
participants
  Complete Response | 0
  Partial Response | 6
  Stable Disease | 16
  Progression of Disease | 27

2. Secondary Outcome: Overall Survival
Description: Overall survival at 18 months post treatment
Time Frame: 18 months after ending treatment
Measure: Number; unit: percentage of participants
Arm/Group | Temozolomide (TMZ)
Number analyzed (Participants) | 49
percentage of participants | 27

3. Secondary Outcome: Duration of Objective Clinical Responses
Description: Duration of Response (Objective Clinical Responses)
Time Frame: 24 weeks after ending treatment
Measure: Median (Full Range); unit: months
Arm/Group | Temozolomide (TMZ)
Number analyzed (Participants) | 6
months | 7.7 [4.3 to 11.1]

ADVERSE EVENTS:
Arm/Group | Temozolomide (TMZ)
Serious Adverse Events (participants affected / at risk) | 7/49
Other Adverse Events (participants affected / at risk) | 14/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide (TMZ) (N=49)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Treatment-related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lymphocyte count decrease (Investigations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide (TMZ) (N=49)
Lymphocyte count decrease (Investigations) | 14 (14)
Anemia (Blood and lymphatic system disorders) | 6 (6)
WBC/Neutropenia (Investigations) | 3 (3)
Nausea/Vomiting (Gastrointestinal disorders) | 8 (8)
Anorexia (Metabolism and nutrition disorders) | 4 (4)
Hyperbilirubinemia (Investigations) | 5 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (7)
Fatigue (General disorders) | 7 (7)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes